CLINICAL TRIAL: NCT00497029
Title: Early Childhood Caries Prevention at a Pediatric Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Minah-1
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2007-07

CONDITIONS: Dental Caries
Keywords: dental caries; early childhood caries; caries prevention; infants
MeSH Terms: conditions — Dental Caries | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluoride varnish
Behavioral: patient education

SUMMARY:
This purpose of this study was to evaluate effectiveness of a risk-based dental caries prevention program conducted by dental personnel at an urban pediatric primary care clinic serving largely low-income residents of Baltimore, Maryland, and to appraise this program as a model for similar urban pediatric settings.

DETAILED DESCRIPTION:
A demonstration caries prevention trial lasting 26 months was conducted with a total of 219 children aged 6 to 27 months of age. The "prevention" group consisting of children 6-15 months of age at their initial visit were compared at the end of the trial with a "comparison" group at their initial visit. The comparison group was 12 months older than the enrollment age of the prevention group (18-27 months) and had not received previous routine professional dental care. Interventions were dental examination and periodic recalls, caries-risk assessments, monitoring of oral mutans streptococci (MS) levels, application of 5.0% sodium fluoride varnish to teeth, dental health counseling to care-givers, referral for dental treatment if indicated and periodic recalls.

Outcome measures were: 1) number of decayed, missing, filled primary tooth surfaces, 2) number of pre-carious lesions, 3) counts of oral MS and 3) care-giver responses to a questionnaire about the child's diet and home care.

Prevention group children at the last recall experienced fewer mean carious dental surfaces (0.1 vs. 1.29, p<0.014) and over 8-fold less MS (p<0.013) than comparison group subjects at the initial visit. The number of precarious lesions, however, were not significantly different. In the absence of carious or precarious lesions, oral levels of MS was a reliable indicator of caries risk status, particularly for low risk subjects (sensitivity, 0.64; specificity, 0.98). Caregiver reports of dietary practices and presence or absence of visible dental plaque also served as caries-risk determinants.

ELIGIBILITY:
Inclusion Criteria:

* children in good health who were dentate and 6-27 months
* a signed informed consent

Exclusion Criteria:

* antibiotic usage within the previous 14 days
* oral topical fluoride administration within the previous 7 days
* previous routine professional dental care

Ages: 6 Months to 27 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2004-06; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
dmfs scores | 12 months

SECONDARY OUTCOMES:
caries-preventive behaviors by care-givers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn E Minah, DDS, PhD, Principal Investigator — Department of Biomedical Sciences, University of Maryland Dental School; Lindsey K Grossman, MD, Study Director — Department of Pediatrics, University of Maryland School of Medicine
Locations (1):
- University of Maryland Medical Center: Pediatric Ambulatory Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Newacheck PW, Hughes DC, Hung YY, Wong S, Stoddard JJ. The unmet health needs of America's children. Pediatrics. 2000 Apr;105(4 Pt 2):989-97. PMID 10742361
- [Background] Gomez SS, Weber AA. Effectiveness of a caries preventive program in pregnant women and new mothers on their offspring. Int J Paediatr Dent. 2001 Mar;11(2):117-22. doi: 10.1046/j.1365-263x.2001.00255.x. PMID 11310134
- [Background] Weintraub JA, Ramos-Gomez F, Jue B, Shain S, Hoover CI, Featherstone JD, Gansky SA. Fluoride varnish efficacy in preventing early childhood caries. J Dent Res. 2006 Feb;85(2):172-6. doi: 10.1177/154405910608500211. PMID 16434737
- [Background] Recommendations for using fluoride to prevent and control dental caries in the United States. Centers for Disease Control and Prevention. MMWR Recomm Rep. 2001 Aug 17;50(RR-14):1-42. PMID 11521913
- [Background] American Dental Association Council on Scientific Affairs. Professionally applied topical fluoride: evidence-based clinical recommendations. J Am Dent Assoc. 2006 Aug;137(8):1151-9. doi: 10.14219/jada.archive.2006.0356. PMID 16873333
- [Background] Rozier RG, Sutton BK, Bawden JW, Haupt K, Slade GD, King RS. Prevention of early childhood caries in North Carolina medical practices: implications for research and practice. J Dent Educ. 2003 Aug;67(8):876-85. PMID 12959161
- [Background] Bader JD, Rozier RG, Lohr KN, Frame PS. Physicians' roles in preventing dental caries in preschool children: a summary of the evidence for the U.S. Preventive Services Task Force. Am J Prev Med. 2004 May;26(4):315-25. doi: 10.1016/j.amepre.2003.12.001. PMID 15110059
- [Background] Douglass JM, Douglass AB, Silk HJ. Infant oral health education for pediatric and family practice residents. Pediatr Dent. 2005 Jul-Aug;27(4):284-91. PMID 16317967
- [Background] Grindefjord M, Dahllof G, Nilsson B, Modeer T. Prediction of dental caries development in 1-year-old children. Caries Res. 1995;29(5):343-8. doi: 10.1159/000262090. PMID 8521434
- [Background] Barsamian-Wunsch P, Park JH, Watson MR, Tinanoff N, Minah GE. Microbiological screening for cariogenic bacteria in children 9 to 36 months of age. Pediatr Dent. 2004 May-Jun;26(3):231-9. PMID 15185804
- [Background] Alaluusua S, Renkonen OV. Streptococcus mutans establishment and dental caries experience in children from 2 to 4 years old. Scand J Dent Res. 1983 Dec;91(6):453-7. doi: 10.1111/j.1600-0722.1983.tb00845.x. PMID 6581521
- [Background] Kohler B, Andreen I, Jonsson B. The earlier the colonization by mutans streptococci, the higher the caries prevalence at 4 years of age. Oral Microbiol Immunol. 1988 Mar;3(1):14-7. doi: 10.1111/j.1399-302x.1988.tb00598.x. No abstract available. PMID 3268743